CLINICAL TRIAL: NCT01568632
Title: A Phase 1 Study of Imetelstat, a Telomerase Inhibitor, in Children With Refractory or Recurrent Solid Tumors and Lymphomas
Brief Title: Imetelstat for Children With Refractory or Recurrent Solid Tumors and Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120091; 12-C-0091
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Dose Limiting Toxicity; Maximum Tolerated Dose; Telomerase Inhibitor; Safety; Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — imetelstat

INTERVENTIONS:
Drug: Imetelstat

SUMMARY:
Background:

- Imetelstat is a cancer treatment drug that may slow or stop tumor growth. It may also prevent tumors from spreading to other parts of the body. Researchers want to see if it can be a safe and effective treatment for children who have solid tumors or lymphoma that have not responded to other treatments.

Objectives:

- To see if imetelstat is a safe and effective treatment for children who have solid tumors or lymphoma that have not responded to other treatments.

Eligibility:

- Children and adolescents between 1 and 21 years of age who have solid tumors or lymphoma that have not responded to other treatments.

Design:

* Participants will be screened with a physical exam, medical history, and imaging studies. Blood and urine samples will also be collected.
* Participants will receive imetelstat on the first and eighth day of a 21-day cycle of treatment.
* Treatment will be monitored with frequent blood tests and imaging studies. Tumor biopsies may also be performed.
* Participants will keep taking the study drugs for up to a total of 18 cycles as long as the disease does not progress and there are no severe side effects....

DETAILED DESCRIPTION:
BACKGROUND:

* Telomerase is an enzyme that plays a critical role in maintaining telomeres, the specialized structures at the end of chromosomes involved in the replication and stability of the chromosome. Inhibition of telomeres causes the length of the telomere to shorten, and the cell becomes either senescent or undergoes apoptosis.
* In vitro and in vivo studies have demonstrated that imetelstat, a telomerase inhibitor, inhibits primary tumor growth and prevents metastases; while six Phase 1 studies in adults have demonstrated reasonable toxicity profiles with hematologic toxicity the primary cause of dose limiting toxicity.
* Objective responses have been observed with repeated dosing when imetelstat was administered in combination with bortezomib to patients with multiple myeloma, with paclitaxel and bevacizumab to patients with advanced breast cancer, and with paclitaxel plus carboplatin in patients with advanced NSCLC.

OBJECTIVES:

Primary Objectives:

* To estimate the maximum tolerated dose (MTD) and/or recommended Phase 2 dose of imetelstat administered as a 2-hour intravenous infusion, weekly X 2, every 21 days, to children with refractory or recurrent solid tumors.
* To define and describe the toxicities of imetelstat administered on this schedule.
* To characterize the pharmacokinetics of imetelstat in children with recurrent or refractory solid tumors.

Secondary Objectives:

- To preliminarily define antitumor effects of imetelstat and to assess the biological activity by assessing telomerase activity, telomere length, hTERT protein, hTERT mRNA and hTR levels in patient PBMNC samples pretreatment and while on treatment, and assess telomerase activity, hTERT expression and hTERT protein, telomere length, hTERT mRNA and hTR levels in patient's pretreatment tumor samples.

ELIGIBILITY:

- Patients > 12 months and less than or equal to 21 years of age with recurrent or refractory solid tumors, including lymphomas, without CNS tumors or known CNS metastases, and with adequate hematologic, hepatic, renal and cardiac status. Must meet safety laboratory testing levels.

DESIGN:

* In this phase I study, the maximum tolerated dose of imetelstat will be determined using a rolling 6 design where a minimum of 2 evaluable patients will be entered at each of 4 dose levels, where imetelstat is administered intravenously over two hours on Day 1 and 8 of a 21-day cycle in children with recurrent or refractory solid tumors, for up to 17 cycles, up to a total duration of therapy of 18 cycles (approximately 12 months).
* Premedication with acetaminophen and diphenhydramine will be administered prior to each dose; anaphylactic precautions should be adhered to, and steroids may be used for symptom control or as premedication after the first dose. Doses subsequent to the first dose may be delayed or withheld for toxicity.

This study will include a required pharmacokinetic component, and one optional PK draw at 48 hours after the first dose (Day 1, Cycle 1). Patients will be asked to participate in optional blood and tissue correlative biology studies. Radiology studies will undergo central radiology review.

- Once MTD has been defined, up to 12 additional patients with relapsed/refractory solid tumors, including

CNS tumors and lymphomas, may be enrolled to acquire additional PK data at the recommended phase 2 dose, attempting to enroll at least 6 patients < 12 years of age. With a maximum number of patients of

45, this study is anticipated to be completed within 22 to 25 months. Up to 5 patients will be enrolled at NCI.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: Patients must be > than 12 months and less than or equal to 21 years of age at the time of study enrollment.
* Diagnosis: Patients with refractory or recurrent solid tumors, including lymphomas, without CNS tumors or known CNS metastases are eligible for the initial dose escalation phase (Part A). Once the MTD or recommended phase 2 dose has been defined, patients with CNS tumors or known CNS metastases may enroll in the expanded cohort (Part B). All patients must have had histologic verification of malignancy at original diagnosis or relapse except patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of CSF or serum tumor markers including alphafetoprotein or beta-HCG.
* Disease Status: Patients must have either measurable or evaluable disease
* Therapeutic Options: Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with anacceptable quality of life.
* Performance Level: Karnofsky greater than or equal to 50% for patients > 16 years of age and Lansky greater than or equal to 50 for patients less than 16 years of age. Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for a minimum of 1 week prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior Therapy

- Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy, immunotherapy, or radiotherapy.

1. Myelosuppressive chemotherapy: Must not have received

   myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
2. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
3. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
4. Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines.
5. Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody.
6. XRT: greater than or equal to 2 weeks for local palliative XRT (small port); : greater than or equal to 24 weeks must have elapsed if prior TBI, craniospinal XRT or if : greater than or equal to 50% radiation of pelvis; greater than or equal to 6 weeks must have elapsed if other substantial BM radiation.
7. Stem Cell Infusion without TBI: No evidence of active graft vs. host disease and : greater than or equal to 12 weeks must have elapsed since transplant or stem cell infusion. Patients with prior allogeneic transplants are not eligible.

Organ Function Requirements

- Adequate Bone Marrow Function Defined as:

1. For patients with solid tumors without known bone marrow involvement:

   - Peripheral absolute neutrophil count (ANC) : greater than or equal to 1000/mm(3)
   * Platelet count : greater than or equal to 100,000/mm(3) (transfusion independent, defined as not receiving platelet transfusions within a 7 day period priorto enrollment)
2. Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts in

   -.a (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity. At least 5 of every cohort of 6 patients with a solid tumor must be evaluable for hematologic toxicity. If dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity.

   - Adequate Renal Function Defined as:
   * Creatinine clearance or radioisotope GFR greater than or equal to 70ml/min/1.73 m(2) or
   * A serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL)

   Male Female

   1 to < 2 years 0.6 0.6

   2 to < 6 years 0.8 0.8

   6 to < 10 years 1 1

   10 to < 13 years 1.2 1.2

   13 to < 16 years 1.5 1.4

   greater than or equal to 16 years1.7 1.4

   - Adequate Liver Function Defined as:

   - Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 x upper limit of normal (ULN) for age

   - SGPT (ALT) less than or equal to 110 U/L. For the purpose of this study, the ULN for

   SGPT is 45 U/L.

   - Serum albumin greater than or equal to 2 g/dL

   Adequate Coagulation Defined as:

   - aPTT < 1.2 x ULN

   Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

   EXCLUSION CRITERIA:

   - Pregnancy or Breast-Feeding

   Pregnant or breast-feeding women will not be entered on this study, because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

   Concomitant Medications

   - Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the prior 7 days are not eligible.

   - Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.

   - Anti-cancer Agents: Patients who are currently receiving other anticancer agents are not eligible.

   - Anti-GVHD or agents to prevent organ rejection post-transplant:

   Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post transplant are not eligible for this trial.
   * Infection: Patients who have an uncontrolled infection are not eligible.
   * Prior or current CNS bleed (Part B): Patients with CNS tumors or known CNS metastases who have imaging evidence of a prior or current CNS hemorrhage on the baseline MRI obtained within 14 days prior to study enrollment are not eligible. Note: The presence of small punctate areas consistent with hemorrhage on ECHO gradient MRI sequences will not exclude patients from participation.
   * Patients with prior allogeneic transplants are not eligible.
   * Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose (MTD) of imetelstat given as a 2-hour IV infusion on D1 and D8 every 21 days.
Define the toxicities and characterize pharmacokinetics

SECONDARY OUTCOMES:
To define antitumor effects and to assess the biological activity by assessing telomerase activity, telomere length, hTERT protein, hTERT mRNA and hTR levels; hTERT expression and protein, telomere length, hTERT mRNAS and hTR levels in tumor.

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Harley CB, Futcher AB, Greider CW. Telomeres shorten during ageing of human fibroblasts. Nature. 1990 May 31;345(6274):458-60. doi: 10.1038/345458a0. PMID 2342578
- [Background] Harley CB. Telomerase is not an oncogene. Oncogene. 2002 Jan 21;21(4):494-502. doi: 10.1038/sj.onc.1205076. PMID 11850774
- [Background] Bosoy D, Peng Y, Mian IS, Lue NF. Conserved N-terminal motifs of telomerase reverse transcriptase required for ribonucleoprotein assembly in vivo. J Biol Chem. 2003 Feb 7;278(6):3882-90. doi: 10.1074/jbc.M210645200. Epub 2002 Nov 27. PMID 12458198